CLINICAL TRIAL: NCT03131323
Title: Nasal Findings in Reactive Airway Diseases
Acronym: nasalfinding
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, lamiaa mahmoud, doctor, Assiut University
Other Study IDs: Assuit universit 17100106
Record Dates: First submitted 2017-04-23; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Reactive Airway Disease; Wheezing
Keywords: delineate the prevalence of abnormal nasal finding in wheezy child
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: • Flexible fiberopticnasopharyngoscope — .
  II- Equipments:
  * Flexible fiberopticnasopharyngoscope, 2.7 mm in diameter and fiberoptic light cable.
  * The camera: fitted with Three-CCD (Charged Couple Device) sensors.
  * A high resolution monitor.
  * A recording unit. III- Positioning:Infants and small children have to be held by a parent or an adult. Older children and adolescents usually tolerate office flexible nasopharyngoscopy once the procedure is explained. If office flexible nasopharyngoscopy failed because the child is not cooperative or if there is excessive secretions, general anesthesia may be required [8].
  IV- Technique: Lubricant gel will be applied to the tip of the endoscope which will be now will be passed along the floor of the nose, between the inferior turbinate and the nasal septum, till it reaches the nasopharynx. Now the entire nose and the nasopharynx could be thoroughly examined and any abnormal findings could be detected and documented.

SUMMARY:
Reactive airway diseases is a common respiratory diseases affecting 1-18% of the population in different countries. It carries a significant burden to children, their families, the healthcare system and the overall community.The purpose of the study is to delineate the prevalence of abnormal nasal finding in wheezy children and evaluate the role of the endoscopic examination of the nose in evaluation and management of a wheezy child.Patients and methods:The study will be conducted as a prospective case series including all children having chest wheezes, aged from two years to eighteen years, attending emergency unit of assuit university children hospital

DETAILED DESCRIPTION:
Reactive airway diseases is a common respiratory diseases affecting 1-18% of the population in different countries. The worldwide increasing incidence of asthma continues to make it a global health problem . It is one of the major causes of hospitalization among children younger than 15 years of age . It carries a significant burden to children, their families, the healthcare system and the overall community. When combined with shortness of breath, chest tightness and/or cough, it is a bronchial asthma .

Pediatric wheeze be triggered by upper respiratory tract infections . The adenoids are a prominent contributor to chronic rhinitis in the pediatric population. Clinical control of chronic rhinosinusitis may be important to optimize the control of difficult-to-treat asthma. However, the relationship between chronic rhinosinusitis and asthma in children remains largely descriptive .

ELIGIBILITY:
Inclusion Criteria:

* All children having chest wheezes, aged from two years to eighteen years, attending emergency unit of Assiut University Pediatric Hospital, during the period 1⁄6∕2017 to 1∕6⁄2018. They will be examined in Otolaryngology Department, Assiut University Hospital

Exclusion Criteria:

* Refusal of endoscopic nasal examination by care givers.and patients with definite diagnosis of wheeze (bronchiolitis,pneumonia)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children aged from 2years to 18 years with recurrent wheezy ches
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
nasal findings in reactive airway diseases | one year
  the prevalence of abnormal nasal finding in wheezy children

IPD SHARING:
Plan to Share IPD: Undecided
children with age group 2years to 18 years will be obtained at the start of the study attenindin to emergency unit